CLINICAL TRIAL: NCT05781984
Title: Role of Surgery in Management of Pineal Region Tumors in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Ibrahim Alghriany, Assistan lecturer of Neurosurgery, Assiut University
Other Study IDs: Pineal Region Tumors
Record Dates: First submitted 2023-03-12; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Brain Tumor
Keywords: pineal region
MeSH Terms: conditions — Brain Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Microsugical Excsosion — Microsurgical excision of pineal region tumor or endoscopic biopsy
  Other Names: Endoscopic Biopsy

SUMMARY:
The aim of this observational study is to learn about the role of surgery with its different approaches and modalities in the management of pineal region tumors in pediatric population.the main question it aims to answer is : How can surgery affect the outcome in children with pineal region tumors ?

ELIGIBILITY:
Inclusion Criteria:

* All patients with pineal region tumors with age less than or equal to 18 years old and fit for surgical intervention

Exclusion Criteria:

* patients with pineal region tumors older than 18 years old
* and pediatric patients younger than 18 years ild and unfit for surgical intervention

Ages: 2 Months to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric population with age of 18 years old or younger diagnosed with pineal region tumor and fit for surgical intervention
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
role of surgery and its effect in improving quality of life in children with pineal region tumors | three years
  evaluation of effect of surgical management with its different approaches in improvement of quality of life and performance status using Karnofsky Performance score (KPS) and radiological imaging till referral to adjuvant therapy

REFERENCES:
- [Background] Choudhry O, Gupta G, Prestigiacomo CJ. On the surgery of the seat of the soul: the pineal gland and the history of its surgical approaches. Neurosurg Clin N Am. 2011 Jul;22(3):321-33, vii. doi: 10.1016/j.nec.2011.04.001. PMID 21801980
- [Background] Li Y, Zhao G, Wang H, Zhu W, Qu L, Li Y, Yu J. Use of 3D-computed tomography angiography for planning the surgical removal of pineal region meningiomas using Poppen's approach: a report of ten cases and a literature review. World J Surg Oncol. 2011 Jun 15;9:64. doi: 10.1186/1477-7819-9-64. PMID 21676231
- [Background] Blakeley JO, Grossman SA. Management of pineal region tumors. Curr Treat Options Oncol. 2006 Nov;7(6):505-16. doi: 10.1007/s11864-006-0025-6. PMID 17032562
- [Background] Mottolese C, Szathmari A, Beuriat PA. Incidence of pineal tumours. A review of the literature. Neurochirurgie. 2015 Apr-Jun;61(2-3):65-9. doi: 10.1016/j.neuchi.2014.01.005. Epub 2014 Aug 10. PMID 25113513
- [Background] Mori Y, Kobayashi T, Hasegawa T, Yoshida K, Kida Y. Stereotactic radiosurgery for pineal and related tumors. Prog Neurol Surg. 2009;23:106-118. doi: 10.1159/000210057. Epub 2009 Mar 23. PMID 19329865
- [Background] Wang P, Mao Q, Wang W, Zhou LX, Liu YH. Gamma knife surgery for pineal region tumors: an alternative strategy for negative pathology. Arq Neuropsiquiatr. 2014 Feb;72(2):129-35. doi: 10.1590/0004-282X20130217. PMID 24604367
- [Background] Behari S, Garg P, Jaiswal S, Nair A, Naval R, Jaiswal AK. Major surgical approaches to the posterior third ventricular region: A pictorial review. J Pediatr Neurosci. 2010 Jul;5(2):97-101. doi: 10.4103/1817-1745.76093. No abstract available. PMID 21559151
- [Background] Poppen JL. The right occipital approach to a pinealoma. J Neurosurg. 1966 Dec;25(6):706-10. doi: 10.3171/jns.1966.25.6.0706. No abstract available. PMID 5925731
- [Background] Dandy WE. EXTIRPATION OF THE PINEAL BODY. J Exp Med. 1915 Aug 1;22(2):237-46. doi: 10.1084/jem.22.2.237. PMID 19867913
- [Background] Morgenstern PF, Souweidane MM. Pineal region tumors: simultaneous endoscopic third ventriculostomy and tumor biopsy. World Neurosurg. 2013 Feb;79(2 Suppl):S18.e9-13. doi: 10.1016/j.wneu.2012.02.020. Epub 2012 Feb 10. PMID 22381843
- [Background] Masina R, Ansaripour A, Benes V, Berhouma M, Choque-Velasquez J, Eide PK, Fedorko S, Fleck S, Hernesniemi J, Koziarski A, Majovsky M, Podgorski A, Schroeder H, Teo C, Unterberg AW, Yeung JT, Kolias A, Santarius T. Surgical treatment of symptomatic pineal cysts without hydrocephalus-meta-analysis of the published literature. Acta Neurochir (Wien). 2022 Jan;164(1):61-77. doi: 10.1007/s00701-021-05054-0. Epub 2021 Dec 2. PMID 34854993